CLINICAL TRIAL: NCT00551473
Title: An Open-Label Study of the Development of Pharmacodynamic Tolerance to 7-days Administration of Lavoltidine 40mg
Brief Title: Open-label Comparison of 24hr Gastric pH on Days 1, 2, 7 With Once-daily Administration of Lavoltidine 40 mg.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LAV110285
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Gastroesophageal Reflux Disease; Reflux, Gastroesophageal
Keywords: pharmacodynamics,; tolerance; H2 antagonist,; AH23844,; lavoltidine,; gastroesophageal reflux disease (GERD), pharmacokinetics,
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lavoltidine

SUMMARY:
Current treatment for gastroesophageal reflux disease(GERD)confirms an unmet need in patients, based on slow onset of action and an inability to provide 24-hour gastric acid suppression. Clinical data on lavoltidine demonstrates a rapid onset of action, high potency, and prolonged duration of effect after single dose. Since tolerance to the class of compounds to which lavoltidine belongs may be dose dependent, the current study is designed to determine if 40mg lavoltdine given for 7days develops tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, from 18-55 years
* Have BMI from 19-30 kg/m2
* do not present with abnormal clinical lab findings
* are able to tolerate a nasogastric pH electrode.

Exclusion Criteria:

* Helicobacter-positive on a C13 urea breath test
* have a baseline median 24-hour gastric pH>3

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05

PRIMARY OUTCOMES:
To determine the degree of pharmacodynamic tolerance following seven days administration of lavoltidine 40mg on gastric pH as assessed by percentage of 24hrs pH>4. | seven days

SECONDARY OUTCOMES:
To determine whether or not significant pharmacodynamic tolerance occurs as early as the second dose of 40mg lavoltidine. Safety and tolerance of seven days administration of lavoltidine 40 mg, in healthy male volunteers. | seven days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, Sydney, New South Wales, Australia